CLINICAL TRIAL: NCT04559308
Title: The Effect of Metformin on Breast Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Collaborators: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Hadeer Mohamed Ehab, Clinical Pharmacy Researcher, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSU
Record Dates: First submitted 2020-08-22; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer
Keywords: Metformin; Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Metformin; Drug Therapy; Doxorubicin; Cyclophosphamide; Paclitaxel

STUDY DESIGN:
Intervention Model Description: The study is an open-labeled, parallel, randomized controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- metformin arm (Experimental): 4 cycles (Doxorubicin+Cyclophosphamide) followed by 12 cycles Paclitaxel+ Metformin (1000 mg twice daily) followed by surgery.
  Interventions: Drug: Metformin; Drug: Chemotherapy
- control arm (Active Comparator): 4 cycles (Doxorubicin+Cyclophosphamide) followed by 12 cycles Paclitaxel followed by surgery.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Metformin — first-line anti-diabetic drug
  Other Names: Glucophage
  Arms: metformin arm
Drug: Chemotherapy — First line neoadjuvant chemotherapy protocol
  Other Names: Doxorubicin; Cyclophosphamide; Paclitaxel

SUMMARY:
Several clinical trials have addressed the promising anticancer effect of metformin on the survival benefits, clinical response, and pathological response of breast cancer patients.

Therefore, this study will assess the anticancer effect of metformin when added to the neoadjuvant chemotherapy protocol of non-diabetic breast cancer patients. In addition to, the impact of metformin addition to the neoadjuvant chemotherapy on the quality of life of breast cancer patients.

DETAILED DESCRIPTION:
This study is conducted to assess the effect of metformin addition to the chemotherapy protocol of non-diabetic breast cancer patients compared to the control group (non-metformin users) in the neoadjuvant setting. Evaluation of the the clinical benefit rate and the rate of pathological complete response will be conducted. In addition, a correlation between the beneficial effect of metformin and the serum concentration of metformin. Also, a comparison in the quality of life between the metformin group and the control group will be evaluated using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ C30) and (EORTC QLQ BR45) questionnaires will be done.

ELIGIBILITY:
Inclusion Criteria:

1. Non-diabetic breast cancer patients, receiving neoadjuvant chemotherapy treatment.
2. Female Age between 18- 65 years.
3. Written informed consent.

Exclusion Criteria:

1. Known hypersensitivity reaction to Metformin.
2. Intolerable Metformin GI complaints.
3. Patients at risk of lactic acidosis.
4. Diabetic breast cancer patients.
5. Body Mass Index < 18.5 (underweight breast cancer patients).
6. Renal impairment, eGFR <45 mL/min/1.73 m².

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female breast cancer patients
Enrollment: 80 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit rate (Tumor size) | 8 months
  Tumor size measured in calipers from baseline till the last cycle of neoadjuvant chemotherapy.

SECONDARY OUTCOMES:
Pathological complete response | 8 months
  The absence of residual invasive cancer on hematoxylin and eosin evaluation of the resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy.
Number of participants with metformin-related adverse events | 8 months
  Safety and tolerability of conventional anti-diabetic dose of metformin use in breast cancer patients.
The effect of metformin on the quality of life of breast cancer patients | 8 months
  A comparison between the metformin arm and the control arm in the change of quality of life from baseline using the European Organization for Research and Treatment of Cancer (EORTC QLQ C30 tools. Scoring of the EORTC QLQ-C30 is performed according to the EORTC scoring manual. After the scoring procedures, all the responses to likert-scale items were linearly transformed to a 0-100 scale. Higher scores for functional scales and the global quality of life scale, indicate better quality of life, while for symptom scales and single items, a higher score indicates a higher severity of the symptoms and worse quality of life.
The effect of metformin on the quality of life of breast cancer patients | 8 months
  A comparison between the metformin arm and the control arm in the change of quality of life from baseline using the European Organization for Research and Treatment of Cancer (EORTC QLQ BR45).Scoring of the EORTC QLQ-Br45 is performed according to the EORTC scoring manual. After the scoring procedures, all the responses to likert-scale items were linearly transformed to a 0-100 scale. Higher scores for functional scales and the global quality of life scale, indicate better quality of life, while for symptom scales and single items, a higher score indicates a higher severity of the symptoms and worse quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A El Berry, Ph.D., Study Director — Beni-Suef University
Locations (1):
- Beni-suef university, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, safety and efficacy criteria, and statistical analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year
Access Criteria: sent by e-mail